CLINICAL TRIAL: NCT00902070
Title: Protocol for Eslax Intravenous Drug Use Investigation
Brief Title: Protocol for Eslax Intravenous Drug Use Investigation (Study P06082)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P06082
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients to whom Eslax has been administered to relax muscles at the time of anesthesia or tracheal intubation
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Normally, for adults, 0.6 mg/kg of rocuronium bromide is intravenously administered to support endotracheal intubation. If additional administration is necessary, 0.1 - 0.2 mg/kg is intravenously administered. In the case of continuous infusion, infusion is initiated at a rate of 7 μg/kg/min. Dosage should be adjusted based on the age or symptom. The upper limit of this drug for the intubation is 0.9 mg/kg.
  Other Names: Eslax

SUMMARY:
The main purpose of this investigation is to collect safety and efficacy information of Eslax Intravenous 25mg/2.5mL and 50mg/5.0mL (hereinafter referred to as "Eslax") in daily clinical settings.

DETAILED DESCRIPTION:
Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Patients to whom Eslax has been administered to relax muscles at the time of anesthesia or tracheal intubation.

Exclusion Criteria:

* Patients with a history of hypersensitivity to Eslax or bromide.
* Patients with myasthenia gravis or myasthenic syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese 3000 patients
Sampling Method: Non-Probability Sample
Enrollment: 3969 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
incidence of adverse events | The standard observation period for a patient is duration of hospital stay (from one week before Eslax administration to one week after administration at a maximum).

SECONDARY OUTCOMES:
intubation score | From administration of Eslax to completion of intubation
intubation completion time | From administration of Eslax to completion of intubation